CLINICAL TRIAL: NCT01147848
Title: A Randomised, Double-blind, Double-dummy, Parallel-group Multicentre Study to Assess Efficacy and Safety of Fluticasone Furoate/GW642444 Inhalation Powder and Fluticasone Propionate/Salmeterol Inhalation Powder in the Treatment of Persistent Asthma in Adults and Adolescents
Brief Title: HZA113091 Efficacy and Safety of Fluticasone Furoate/Vilanterol (GW642444) in Adults and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113091
Record Dates: First submitted 2010-05-27; First posted 2010-06-22 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Salmeterol; fluticasone furoate; Vilanterol; fluticasone propionate; GW642444
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone furoate/Vilanterol (GW642444) (Experimental): Fluticasone furoate/vilanterol inhalation powder once daily + placebo inhalation powder twice daily for 24 weeks
  Interventions: Drug: Fluticasone furoate/Vilanterol Inhalation Powder; Drug: Placebo (2)
- Fluticasone propionate/salmeterol (Active Comparator): Fluticasone propionate/salmeterol inhalation powder twice daily + placebo inhalation powder once daily for 24 weeks
  Interventions: Drug: Fluticasone propionate/salmeterol Inhalation Powder; Drug: Placebo (1)

INTERVENTIONS:
Drug: Fluticasone furoate/Vilanterol Inhalation Powder — Fluticasone furoate/Vilanterol Inhalation Powder inhaled orally once daily for 24 weeks
  Arms: Fluticasone furoate/Vilanterol (GW642444)
Drug: Fluticasone propionate/salmeterol Inhalation Powder — Fluticasone propionate/salmeterol Inhalation Powder inhaled orally twice daily for 24 weeks
  Arms: Fluticasone propionate/salmeterol
Drug: Placebo (1) — Inhalation powder inhaled orally once daily for 24 weeks
  Arms: Fluticasone propionate/salmeterol
Drug: Placebo (2) — Inhalation powder inhaled orally twice daily for 24 weeks
  Arms: Fluticasone furoate/Vilanterol (GW642444)

SUMMARY:
The purpose of the study is to compare the efficacy and safety of fluticasone furoate/vilanterol (GW642444) inhalation powder administered once daily with fluticasone propionate/salmeterol administered twice daily in adolescent and adult subjects 12 years of age and older with persistent bronchial asthma over a 24-week period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma
* Reversibility of at least 12% and at least 200mLs within 10-40 minutes following 2-4 inhalations of albuterol
* FEV1 of 40-85% predicted normal
* Currently using inhaled corticosteroid therapy

Exclusion Criteria:

* History of life-threatening asthma within previous 5 years (requiring intubation and/or was associated with hypercapnoea, respiratory arrest or hypoxic seizures)
* Respiratory infection or oral candidiasis
* Asthma exacerbation requiring oral corticosteroids or that resulted in overnight hospitalisation requiring additional asthma treatment
* Uncontrolled disease or clinical abnormality
* Allergies
* Taking another investigational medication or prohibited medication
* Night shift workers
* Current smokers or subjects with smoking history of at least 10 pack years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (55):
- United States (24):
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
- Argentina (7):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, Paraná, Entre Ríos Province
  - GSK Investigational Site, Mendoza, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán
- Chile (5):
  - GSK Investigational Site, Rancagua, Reg Del Libert Bern Ohiggins
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Netherlands (8):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Dordrecht
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Veldhoven
- Philippines (6):
  - GSK Investigational Site, Cabanatuan City, Nueva Ecija
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Dasmariñas, Cavite
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Marilao, Bulacan
  - GSK Investigational Site, Quezon City
- South Korea (5):
  - GSK Investigational Site, Cheongju, Chungcheongbuk-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Woodcock A, Bleecker ER, Lotvall J, O'Byrne PM, Bateman ED, Medley H, Ellsworth A, Jacques L, Busse WW. Efficacy and safety of fluticasone furoate/vilanterol compared with fluticasone propionate/salmeterol combination in adult and adolescent patients with persistent asthma: a randomized trial. Chest. 2013 Oct;144(4):1222-1229. doi: 10.1378/chest.13-0178. PMID 23846316
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113091 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluticasone Propionate 250 µg BID: Participants received Fluticasone Propionate 250 micrograms (µg) twice a day (BID) and salbutamol/albuterol as required to control symptoms.
- Fluticasone Furoate/Vilanterol 100/25 µg OD: Participants received Fluticasone Furoate (FF)/Vilanterol (VI) 100/25 µg once daily (OD) in the evening, plus placebo inhalation powder twice daily (BID; in the morning and evening) for a period of 24 weeks.
- Fluticasone Propionate/Salmeterol 250/50 µg BID: Participants received Fluticasone Propionate (FP)/Salmeterol 250/50 µg inhalation powder BID (in the morning and evening), plus placebo inhalation powder OD in the evening for a period of 24 weeks.
Period: Run-in Period
Arm/Group | Fluticasone Propionate 250 µg BID | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Started | 1564 | 0 | 0
Completed | 806 | 0 | 0
Not Completed | 758 | 0 | 0
Not completed — Screen Failure | 623 | 0 | 0
Not completed — Run-in Failure | 135 | 0 | 0
Period: Randomized Phase
Arm/Group | Fluticasone Propionate 250 µg BID | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Started | 0 | 403 | 403
Completed | 0 | 358 | 357
Not Completed | 0 | 45 | 46
Not completed — Adverse Event | 0 | 6 | 8
Not completed — Lack of Efficacy | 0 | 20 | 11
Not completed — Protocol Violation | 0 | 7 | 10
Not completed — Lost to Follow-up | 0 | 5 | 7
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID | Total
Number analyzed (Participants) | 403 | 403 | 806
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.8 (15.86) | 41.9 (16.90) | 42.8 (16.41)
Gender [Count of Participants; unit: Participants]
  Female | 244 | 245 | 489
  Male | 159 | 158 | 317
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 36 | 43 | 79
  Asian - Central/South Asian Heritage | 1 | 0 | 1
  Asian - East Asian Heritage | 40 | 46 | 86
  Asian - Japanese Heritage | 1 | 0 | 1
  Asian - South East Asian Heritage | 81 | 79 | 160
  Asian - Mixed Race | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White - Arabic/North African Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 241 | 232 | 473
  Mixed Race | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weighted-mean 24 Hour Serial FEV1 on Day 168/Week 24
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. The weighted mean was calculated from the pre-dose FEV1 and post-dose FEV1 measurements at 5, 15, and 30 minutes (min) and at 1, 2, 3, 4, 11, 12, 12.5, 13, 14, 16, 20, 23, and 24 hours, respectively, on Day 168/Week 24. Change from Baseline was calculated as the weighted mean of the 24-hour serial FEV1 measures on Day 168/Week 24 minus the Baseline value. Baseline was the pre-dose measurement on Day 1. Analysis was performed using analysis of covariance (ANCOVA) with covariates of Baseline FEV1, region, sex, age, and treatment.
Time Frame: Baseline and Day 168/Week 24
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least 1 dose of double-blind medication. Randomized participants were assumed to have received double-blind medication unless definitive evidence to the contrary existed. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 352 | 347
Liters | 0.341 (0.0184) | 0.377 (0.0185)
Statistical Analysis 1: Comparison: Fluticasone Furoate/Vilanterol 100/25 µg OD vs Fluticasone Propionate/Salmeterol 250/50 µg BID; Test type: Superiority or Other; p = 0.162, ANCOVA; Least Squares Mean Difference = -0.037, 95% CI 2-sided [-0.088 to 0.015] — Analysis was performed using ANCOVA with covariates of Baseline FEV1, region, sex, age, and treatment

2. Secondary Outcome: Serial FEV1 (0-24 Hours)
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second . The pre-dose FEV1 assessment and the individual serial FEV1 assessments at Day 168/Week 24 at the indicated time points (pre-dose, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 11 hours, 12 hours, 12.5 hours, 13 hours, 14 hours, 16 hours, 20 hours, 23 hours, and 24 hour s) were summarized.
Time Frame: Day 168
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 359 | 354
Liters
  Pre-dose, n=359,353 | 0.304 (0.3575) | 0.323 (0.4289)
  5 minutes, n=356, 344 | 0.320 (0.3573) | 0.339 (0.4146)
  15 minutes, n=355, 347 | 0.323 (0.3565) | 0.354 (0.4054)
  30 minutes, n=357, 351 | 0.339 (0.3614) | 0.366 (0.4184)
  1 hour, n=358, 353 | 0.344 (0.3760) | 0.390 (0.4227)
  2 hours, n=359, 353 | 0.362 (0.3749) | 0.409 (0.4204)
  3 hours, n=357, 353 | 0.373 (0.3764) | 0.419 (0.4173)
  4 hours, n=357, 354 | 0.356 (0.3695) | 0.417 (0.4254)
  11 hours, n=359, 347 | 0.305 (0.3761) | 0.319 (0.4099)
  12 hours, n=356, 354 | 0.330 (0.3691) | 0.338 (0.4142)
  12.5 hours, n=357, 352 | 0.330 (0.3682) | 0.380 (0.4117)
  13 hours, n=354, 354 | 0.343 (0.3602) | 0.396 (0.4139)
  14 hours, n=356, 353 | 0.357 (0.3643) | 0.426 (0.4201)
  16 hours, n=354, 350 | 0.351 (0.3672) | 0.419 (0.4152)
  20 hours, n=355, 352 | 0.321 (0.3757) | 0.376 (0.4150)
  23 hours, n=354, 353 | 0.310 (0.3814) | 0.344 (0.4141)
  24 hours, n=354, 354 | 0.304 (0.3725) | 0.340 (0.4032)

3. Secondary Outcome: Number of Participants With the Indicated Time to Onset of Bronchodilator Effect at Day 1
Description: Time to onset of bronchodilator effect at Day 1 is defined as the actual time during the 4-hour serial FEV1 (the maximal amount of air that can be forcefully exhaled in one second) measurements that the participant first meets or exceeds a 12% and 200 mL increase over Baseline and was derived at Day 1 only. Time to onset was calculated over 0 to 4 hours (5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, and 4 hours) post-dose. Participants who never exceeded a 12% and 200 mL increase over Baseline were censored at the actual time of their last FEV1 measurement.
Time Frame: Baseline to Day 1
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Number; unit: participants
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 400 | 401
participants
  5 minutes | 100 | 85
  15 minutes | 41 | 51
  30 minutes | 40 | 55
  1 hour | 32 | 39
  2 hours | 19 | 29
  3 hours | 17 | 12
  4 hours | 11 | 12
  Censored | 140 | 118

4. Secondary Outcome: Change From Baseline in Weighted Mean Serial FEV1 Over 0-4 Hours Post First Dose (at Randomization)
Description: The weighted mean serial FEV1 (the maximal amount of air that can be forcefully exhaled in one second) over 0-4 hours post-dose at Baseline was derived using actual times and using the pre-dose assessment as the 0 hour measurement. Change from Baseline was calculated as the weighted mean of the 4-hour serial FEV1 measures on Day 1 minus the Baseline value. Baseline was the pre-dose measurement on Day 1. Analysis was performed using ANCOVA with covariates of Baseline FEV1, region, sex, age, and treatment.
Time Frame: Baseline and Randomization
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- FFluticasone Furoate/Vilanterol 100/25 µg OD: Participants received Fluticasone Furoate (FF)/Vilanterol (VI) 100/25 µg once daily (OD) in the evening, plus placebo inhalation powder twice daily (BID; in the morning and evening) for a period of 24 weeks.
Arm/Group | FFluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 398 | 398
Liters | 0.316 (0.0149) | 0.346 (0.0149)

5. Secondary Outcome: Change From Baseline in Weighted Mean Serial FEV1 Over 0-4 Hours at Day 168
Description: The weighted mean serial FEV1 (the maximal amount of air that can be forcefully exhaled in one second) over 0-4 hours post-dose at Baseline and Day 168 was derived using actual times and using the pre-dose assessment as the 0 hour measurement. Change from Baseline was calculated as the weighted mean of the 4-hour serial FEV1 measures on Day 168/Week 24 minus the Baseline value. Baseline was the pre-dose measurement on Day 1. Analysis was performed using ANCOVA with covariates of Baseline FEV1, region, sex, age, and treatment.
Time Frame: Baseline and Day 168
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 356 | 347
Liters | 0.360 (0.0184) | 0.394 (0.0186)

6. Secondary Outcome: Number of Participants Obtaining a >=12% and >=200 mL Increase From Baseline in FEV1
Description: The number of participants obtaining a >=12% and >=200 mL increase from Baseline in FEV1 (the maximal amount of air that can be forcefully exhaled in one second) was evaluated at 12-hours post-dose and at 24-hours post-dose on Day 168.
Time Frame: Baseline and Day 168
Population: ITT Population. Only those participants available at the indicated time points were assessed.
Measure: Number; unit: participants
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 356 | 354
participants
  12 hours post-dose, n=356,354 | 199 | 178
  24 hours post-dose, n=354, 354 | 181 | 176

7. Secondary Outcome: Change From Baseline in Trough FEV1 at Day 168
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second . Trough FEV1 is defined as the pre-dose measurement on Day 168/Week 24. Any missing data at Day 168/Week 24 was imputed using the last observation carried forward (LOCF). Baseline was the pre-dose measurement on Day 1. Change from Baseline was calculated as the pre-dose measurement on Day 168/Week 24 minus the Baseline value.
Time Frame: Baseline and Day 168
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 397 | 389
Liters | 0.281 (0.0191) | 0.300 (0.0193)

8. Other Pre Specified Outcome: Baseline FEV1 by Completion Status
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second . Baseline is defined as the mean of the two assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1.
Time Frame: Baseline
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 401 | 401
Liters
  All Participants, n=401, 401 | 2.011 (0.6389) | 2.048 (0.6246)
  Completers, n=359, 355 | 2.013 (0.6530) | 2.043 (0.6378)
  Withdrawals, n=42, 46 | 1.996 (0.5081) | 2.091 (0.5145)

9. Other Pre Specified Outcome: Change From Baseline in Asthma Control Test (ACT) Scores at Day 168
Description: The ACT is a 5-item questionnaire developed as a measure of the participant's asthma control. Questions are designed to be self-completed by the participant and include the following: In the past 4 weeks, "How much of the time did your asthma keep you from getting as much done at work, school or at home?", "How often have you had shortness of breath?", "How often did your asthma symptoms wake you up at night or earlier than usual in the morning?", "How often have you used your rescue inhaler or nebulizer medication (such as albuterol)?" and "How would you rate your asthma control"? The ACT total score is defined as the sum of the scores from all 5 questions, provided all questions have been answered; thus, the total score ranges from 5 (poor control of asthma) to 25 (complete control of asthma). A score of 20 or higher indicates well-controlled asthma. Change from Baseline was calculated as the Day 168 value minus the Baseline value.
Time Frame: Baseline and Day 168
Population: ITT Population. Only those participants available at the indicated time point were assessed. Analysis was performed using ANCOVA with covariates of Baseline total ACT score, country, sex, age, and treatment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 354 | 348
Scores on a scale | 2.3 (0.16) | 2.0 (0.16)

10. Other Pre Specified Outcome: Number of Healthcare Contacts Related to Asthma or the Treatment of Asthma From Baseline to Day 168
Description: All unscheduled asthma-related visits to a physician's office, visits to urgent care, visits to the emergency department, and hospitalizations (to the general ward [GW] or the intensive care unit [ICU]) that were associated with asthma exacerbations were recorded.
Time Frame: Baseline to Day 168
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Mean (Standard Deviation); unit: visits per participant
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 403 | 403
visits per participant
  Number of Home Visits during the Day | 0.0 (0.0) | 0.0 (0.05)
  Number of Home Visits during the Night | 0.0 (0.0) | 0.0 (0.0)
  Number of Physician Office/Practice Visits | 0.0 (0.29) | 0.0 (0.18)
  Number of Urgent Care/Outpatient Clinic Visits | 0.0 (0.05) | 0.0 (0.05)
  Number of Emergency Room Visits | 0.0 (0.15) | 0.0 (0.14)
  Number of Inpatient Hospitalization (ICU) Days | 0.0 (0.00) | 0.0 (0.0)
  Number of Inpatient Hospitalization (GW) Days | 0.0 (0.20) | 0.0 (0.39)

11. Other Pre Specified Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Total Score for Participants 12 Years of Age and Older (AQLQ + 12)
Description: The AQLQ is a disease-specific, self-administered quality of life (QOL) questionnaire developed to evaluate the impact of asthma treatments on the QOL of asthma sufferers. The AQLQ contains 32 items in four domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items), and environmental stimuli (4 items). The response format consists of a 7-point scale: a value of 1 indicates "total impairment"; a value of 7 indicates "no impairment." The AQLQ total score is defined as the average of the scores from all 32 questions, provided at least 90% of the questions have been answered; thus, the total score ranges from 1 (indicates "total impairment") to 7 (indicates "no impairment"). Change from Baseline was calculated as the Day 168 value minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline total AQLQ score, country, sex, age, and treatment.
Time Frame: Baseline and Day 168
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 342 | 335
Scores on a scale | 0.46 (0.043) | 0.37 (0.043)

12. Other Pre Specified Outcome: Percentage of Participants With "No Problems" in the EQ-5D Descriptive System Dimensions at Day 168/Week 24
Description: The EQ-5D is a standardized, 2-part, self-assessment instrument, designed for self-completion, used to measure health outcome. The first part consists of 5 items covering 5 dimensions (mobility, self care, usual activities, pain/discomfort, and anxiety/depression). Each dimension is measured by a three-point Likert scale (1=no problems, 2=some problems and 3=severe problems). Respondents are asked to choose one level that reflects their "own health state today" for each of the five dimensions.
Time Frame: Day 168/Week 24
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Number; unit: percentage of participants
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 403 | 403
percentage of participants
  Mobility | 86 | 84
  Self care | 98 | 98
  Usual activities | 86 | 82
  Pain/Discomfort | 70 | 66
  Anxiety/Depression | 78 | 81

13. Other Pre Specified Outcome: Change From Baseline in EQ-5D Visual Analog Scale (VAS) Score at Day 168
Description: The EQ-5D is a standardized, 2-part, self-assessment instrument, designed for self-completion, used to measure health outcome. The first part consists of 5 items covering 5 dimensions (mobility, self care, usual activities, pain/discomfort, and anxiety/depression). The second part is a 20 centimeter VAS that has endpoints labelled "best imaginable health state" and "worst imaginable health state" anchored at 100 and 0, respectively. Participants were asked to indicate how they rate their own health by drawing a line from an anchor box to that point on the EQ-VAS that best represents their own health on that day. Analysis was performed using ANCOVA with covariates of Baseline VAS score, country, sex, age, and treatment.
Time Frame: Baseline and Day 168
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 343 | 349
scores on a scale | 5.5 (0.60) | 4.1 (0.60)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of the study medication until Follow-up (up to 544 days).
Description: All AEs and SAEs were followed until resolution, until the condition stabilized, until the event was otherwise explained, or until the participant was lost to follow-up.
Arm/Group | Fluticasone Furoate/Vilanterol 100/25 µg OD | Fluticasone Propionate/Salmeterol 250/50 µg BID
Serious Adverse Events (participants affected / at risk) | 4/403 | 5/403
Other Adverse Events (participants affected / at risk) | 110/403 | 106/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Furoate/Vilanterol 100/25 µg OD (N=403) | Fluticasone Propionate/Salmeterol 250/50 µg BID (N=403)
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Furoate/Vilanterol 100/25 µg OD (N=403) | Fluticasone Propionate/Salmeterol 250/50 µg BID (N=403)
Nasopharyngitis (Infections and infestations) | 46 | 46
Upper respiratory tract infection (Infections and infestations) | 25 | 16
Headache (Nervous system disorders) | 34 | 41
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 13
Pyrexia (General disorders) | 13 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.